CLINICAL TRIAL: NCT02445586
Title: A Phase IV, Multicenter, Open-Label, Single-Arm Study of Pertuzumab (in Combination With Trastuzumab and Docetaxel) in First Line Treatment of Indian Patients With HER2-Positive Advanced (Metastatic or Locally Recurrent) Breast Cancer
Brief Title: Safety Study of Pertuzumab (in Combination With Trastuzumab and Docetaxel) in Indian Participants With Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML29282
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pertuzumab in Combination with Trastuzumab and Docetaxel (Experimental): Participants will receive pertuzumab in combination with trastuzumab and docetaxel every 3 weeks until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: Docetaxel; Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Docetaxel — Participants will receive docetaxel in line with locally approved Prescribing Information. After Cycle 6 (cycle length = 21 days), continuation of docetaxel treatment will be at the discretion of the investigator. Docetaxel will be administered after pertuzumab and trastuzumab.
Drug: Pertuzumab — Participants will receive pertuzumab at an initial dose of 840 milligrams (mg) as a 60-minute intravenous infusion on Cycle 1 Day 1 (cycle length = 21 days), followed by every 3 weeks at a dose of 420 mg as a 30 to 60-minute intravenous infusion until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Other Names: Perjeta®
Drug: Trastuzumab — Participants will receive trastuzumab at an initial dose of 8 milligrams per kilogram (mg/kg) as a 90-minute intravenous infusion on Cycle 1 Day 1 (cycle length = 21 days), followed by every 3 weeks at a dose of 6 mg/kg as a 30 to 90-minute intravenous infusion until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Other Names: Herceptin®; Herclon®

SUMMARY:
This is a Phase 4, single-arm, open-label, multicenter study to assess the safety and efficacy of pertuzumab in combination with trastuzumab and docetaxel for the treatment of participants with human epidermal growth factor receptor 2 (HER2)-positive advanced (locally recurrent, unresectable, or metastatic) breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* For women of childbearing potential and men with partners of childbearing potential, agreement to use a highly-effective non-hormonal form of contraception or two effective forms of non-hormonal contraception by the participant and/or partner
* Histologically or cytologically confirmed and documented adenocarcinoma of the breast with metastatic or locally recurrent disease not amenable to curative resection; participants with measurable and/or non-measurable disease are eligible
* Known and documented HER2-positive
* Known and documented LVEF of at least 50 percent (%)
* Adequate organ function
* A negative serum beta-human chorionic gonadotropin (beta-HCG) test for women of childbearing potential (premenopausal, or less than [<] 12 months of amenorrhea post-menopause, and women who have not undergone surgical sterilization [absence of ovaries and/or uterus]) within 7 days prior to the first dose of study treatment with the result available prior to first dosing

Exclusion Criteria:

* Previous systemic non-hormonal anti-cancer therapy for the metastatic or locally recurrent disease
* Pregnant or lactating women
* Current clinical or radiographic evidence of central nervous system (CNS) metastases
* Disease progression while receiving or within 12 months of completion of trastuzumab and/or lapatinib treatment in the adjuvant or neo-adjuvant setting
* History of LVEF decline to below 50% during or after prior trastuzumab adjuvant or neo-adjuvant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Kukreja, MD, Study Director — Roche Products (India) Pvt. Ltd.
Locations (9):
- India (9):
  - Tata Memorial Hospital; Dept of Medical Oncology, Mumbai, Maharashtra
  - Kokilaben Dhirubhai Ambani Hospital & Medical Research Institute, Mumbai, Maharashtra
  - Jehangir Clinical Development Centre Pvt. Ltd; Cancer Research Room, Pune, Maharashtra
  - Rajiv Gandhi Cancer Institute & Research Center, New Delhi, National Capital Territory of Delhi
  - Christian Medical College & Hospital; Medicine, Vellore, Tamil Nadu
  - Indo-American Cancer Hospital & Research Center, Hyderabad, Telangana
  - TATA Medical Centre; Medical Oncology, Kolkata, West Bengal
  - M S Ramaiah Memorial Hospital, Bangalore
  - MAX Balaji Hospital, Delhi

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Started (Intent-to-Treat (ITT) Population) | 52
Received at Least One Dose of Study Drug (Safety Population) | 52
Completed | 13
Not Completed | 39
Not completed — Death | 14
Not completed — Withdrawal by Subject | 13
Not completed — Disease Progression | 10
Not completed — Protocol Violation | 1
Not completed — Medical Condition | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 52
  Ethnicity: Indian Subcontinent | 52
Diagnosis of Metastatic or Locally Recurrent Breast Cancer [Count of Participants; unit: Participants]
  Metastatic | 52
  Locally Recurrent | 0
Histological Grade of Breast Cancer [Count of Participants; unit: Participants]
  Well Differentiated | 14
  Moderately Differentiated | 16
  Poorly Differentiated | 11
  Anaplastic | 0
  Unknown | 11
Breast Cancer Subtype by Histology [Count of Participants; unit: Participants]
  Ductal | 47
  Lobular | 0
  Other | 5
Presence or Absence of Ductal Carcinoma In Situ (DCIS) [Count of Participants; unit: Participants]
  DCIS Present | 22
  DCIS Absent | 29
  DCIS Assessment Missing | 1
HER2-Positive Breast Cancer Confirmation Method [Count of Participants; unit: Participants] — The human epidermal growth factor receptor 2 (HER2) positive status of each participant's breast cancer was confirmed either by documented evidence from previous testing or by fixed tissue blocks of primary and/or metastatic tumors locally assessed according to institutional criteria and routine clinical practice using immunohistochemistry (IHC), in situ hybridization (ISH), or both methods.
  Participants
    Immunohistochemistry (IHC) | 31
    In Situ Hybridization (ISH) | 1
    Both IHC and ISH | 20
HER2 Expression Score by IHC [Count of Participants; unit: Participants] — The immunohistochemistry (IHC) test measures the amount of human epidermal growth factor receptor 2 (HER2) protein on the surface of cells in a breast cancer tissue sample. A score from 0 to 3+ is assigned with the following significance: a score of 0 or 1+ is considered HER2 negative; a score of 2+ is considered borderline; and a score of 3+ is considered HER2 positive.
  Participants
    0 | 0
    1+ | 0
    2+ | 4
    3+ | 47
    Assessment Missing | 1
HER2 Expression Score by ISH [Count of Participants; unit: Participants] — The in situ hybridization (ISH) test measures human epidermal growth factor receptor 2 (HER2) gene amplification in the DNA of cells from a breast cancer tissue sample and is scored as negative (non-amplified) or positive (amplified).
  Participants
    Negative (Non-Amplified) | 1
    Positive (Amplified) | 20
    Not Assessed by ISH | 31
Hormone Receptor Status (Positive or Negative) [Count of Participants; unit: Participants] — The expression of estrogen and progesterone receptors in metastatic tumors were assessed for positive or negative status.
  Participants
    Estrogen Receptor: Positive | 21
    Estrogen Receptor: Negative | 31
    Progesterone Receptor: Positive | 18
    Progesterone Receptor: Negative | 34
Any Previous Therapy for Breast Cancer [Count of Participants; unit: Participants]
  Yes | 19
  No | 33

OUTCOME MEASURES:

1. Primary Outcome: Overall Number of Participants by the Number of Serious Adverse Events Reported Per Participant
Description: The number of participants with serious adverse events was counted in the four following categories for number of events reported per participant: greater than or equal to (≥) 1, 1, greater than (>) 1, or 0 serious adverse events. Participants with multiple occurrences of events (the ≥1 and >1 serious adverse event categories) were only counted once per category.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  ≥1 Serious Adverse Event | 31
  1 Serious Adverse Event | 17
  >1 Serious Adverse Events | 14
  0 Serious Adverse Events | 21

2. Primary Outcome: Overall Number of Participants With Serious Adverse Events by Severity (Initial and Most Extreme), According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (NCI CTCAE v4.03)
Description: The number of participants with serious adverse events was counted by the initial and most extreme levels of severity of the adverse event, assessed as Grades 1-5 according to NCI CTCAE v4.03. Any adverse event not specifically listed in NCI CTCAE v4.03 was assessed according to the following grades of severity: Grade 1 is mild; Grade 2 is moderate; Grade 3 is severe or medically significant; Grade 4 is life-threatening or urgent intervention indicated; and Grade 5 is death related to adverse event. The terms "severe" and "serious" are not synonymous. Severity refers to the intensity of an adverse event. The seriousness of an adverse event is based on whether it meets any of the criteria set out in the protocol's definition of a serious adverse event. Severity and seriousness were independently assessed for each adverse event. Participants with multiple occurrences of serious adverse events of the same severity were only counted once per severity category.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population; the number analyzed in each category represents the number of participants with at least one serious adverse event (denominator).
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Initial Severity - Grade 1: number analyzed (Participants) | 31
  Initial Severity - Grade 1 | 1
  Initial Severity - Grade 2: number analyzed (Participants) | 31
  Initial Severity - Grade 2 | 4
  Initial Severity - Grade 3: number analyzed (Participants) | 31
  Initial Severity - Grade 3 | 15
  Initial Severity - Grade 4: number analyzed (Participants) | 31
  Initial Severity - Grade 4 | 7
  Initial Severity - Grade 5: number analyzed (Participants) | 31
  Initial Severity - Grade 5 | 14
  Most Extreme Severity - Grade 1: number analyzed (Participants) | 31
  Most Extreme Severity - Grade 1 | 1
  Most Extreme Severity - Grade 2: number analyzed (Participants) | 31
  Most Extreme Severity - Grade 2 | 3
  Most Extreme Severity - Grade 3: number analyzed (Participants) | 31
  Most Extreme Severity - Grade 3 | 16
  Most Extreme Severity - Grade 4: number analyzed (Participants) | 31
  Most Extreme Severity - Grade 4 | 7
  Most Extreme Severity - Grade 5: number analyzed (Participants) | 31
  Most Extreme Severity - Grade 5 | 15

3. Primary Outcome: Number of Participants With Serious Adverse Events Related to Docetaxel
Description: The number of participants with serious adverse events was counted for any serious adverse event that was related to study treatment with docetaxel, in the investigator's judgment. Adverse events (AEs) were encoded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 21.1. More than one serious adverse event may have been reported per participant. Participants with multiple occurrences of the same serious adverse event were only counted once per preferred term.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Any Serious AEs Related to Docetaxel | 15
  Diarrhoea | 5
  Left ventricular dysfunction | 2
  Fatigue | 2
  Sinus tachycardia | 1
  Abdominal pain | 1
  Febrile neutropenia | 1
  Enteritis | 1
  Salivary hypersecretion | 1
  Stomatitis | 1
  Vomiting | 1
  Pyrexia | 1
  Device related sepsis | 1
  Septic shock | 1
  Infusion related reaction | 1
  Rash | 1

4. Primary Outcome: Number of Participants With Serious Adverse Events Related to Pertuzumab
Description: The number of participants with serious adverse events was counted for any serious adverse event that was related to study treatment with pertuzumab, in the investigator's judgment. Adverse events (AEs) were encoded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 21.1. More than one serious adverse event may have been reported per participant. Participants with multiple occurrences of the same serious adverse event were only counted once per preferred term.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Any Serious AEs Related to Pertuzumab | 13
  Diarrhoea | 4
  Ejection fraction decreased | 3
  Left ventricular dysfunction | 2
  Sinus tachycardia | 1
  Abdominal pain | 1
  Enteritis | 1
  Stomatitis | 1
  Fatigue | 1
  Pyrexia | 1
  Gastroenteritis | 1
  Dyspnoea | 1
  Rash | 1
  Shock | 1

5. Primary Outcome: Number of Participants With Serious Adverse Events Related to Trastuzumab
Description: The number of participants with serious adverse events was counted for any serious adverse event that was related to study treatment with trastuzumab, in the investigator's judgment. Adverse events (AEs) were encoded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 21.1. More than one serious adverse event may have been reported per participant. Participants with multiple occurrences of the same serious adverse event were only counted once per preferred term.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Any Serious AEs Related to Trastuzumab | 10
  Ejection fraction decreased | 3
  Left ventricular dysfunction | 2
  Diarrhoea | 2
  Enteritis | 1
  Fatigue | 1
  Pyrexia | 1
  Sinus tachycardia | 1
  Rash | 1
  Shock | 1

6. Primary Outcome: Overall Number of Participants With Serious Adverse Events by Action Taken With Study Drug
Description: The number of participants with serious adverse events was counted by the type of action taken with the study drug (docetaxel, pertuzumab, and trastuzumab) in response to the adverse event in the three following categories: infusion reduced, temporarily interrupted, or permanently discontinued. More than one serious adverse event may have been reported per participant. Participants with multiple occurrences of serious adverse events that required the same action to be taken with the study drug were only counted once per category.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population; the number analyzed represents participants with at least one serious adverse event (denominator).
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Infusion of Docetaxel Reduced: number analyzed (Participants) | 31
  Infusion of Docetaxel Reduced | 0
  Infusion of Docetaxel Temporarily Interrupted: number analyzed (Participants) | 31
  Infusion of Docetaxel Temporarily Interrupted | 1
  Infusion of Docetaxel Permanently Discontinued: number analyzed (Participants) | 31
  Infusion of Docetaxel Permanently Discontinued | 1
  Infusion of Pertuzumab Reduced: number analyzed (Participants) | 31
  Infusion of Pertuzumab Reduced | 0
  Infusion of Pertuzumab Temporarily Interrupted: number analyzed (Participants) | 31
  Infusion of Pertuzumab Temporarily Interrupted | 3
  Infusion of Pertuzumab Permanently Discontinued: number analyzed (Participants) | 31
  Infusion of Pertuzumab Permanently Discontinued | 4
  Infusion of Trastuzumab Reduced: number analyzed (Participants) | 31
  Infusion of Trastuzumab Reduced | 0
  Infusion of Trastuzumab Temporarily Interrupted: number analyzed (Participants) | 31
  Infusion of Trastuzumab Temporarily Interrupted | 3
  Infusion of Trastuzumab Permanently Discontinued: number analyzed (Participants) | 31
  Infusion of Trastuzumab Permanently Discontinued | 5

7. Primary Outcome: Overall Number of Participants With Serious Adverse Events by Event Outcome
Description: The number of participants with serious adverse events was counted by the event outcome in the six following categories: fatal, recovered/resolved, recovered/resolved with sequelae, recovering/resolving, not recovered/not resolved, or unknown. More than one serious adverse event may have been reported per participant. Participants with multiple occurrences of serious adverse events with the same outcome were only counted once per category.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population; the number analyzed represents participants with at least one serious adverse event (denominator).
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Fatal: number analyzed (Participants) | 31
  Fatal | 15
  Recovered / Resolved: number analyzed (Participants) | 31
  Recovered / Resolved | 18
  Recovered / Resolved with Sequelae: number analyzed (Participants) | 31
  Recovered / Resolved with Sequelae | 1
  Recovering / Resolving: number analyzed (Participants) | 31
  Recovering / Resolving | 3
  Not Recovered / Not Resolved: number analyzed (Participants) | 31
  Not Recovered / Not Resolved | 2
  Unknown: number analyzed (Participants) | 31
  Unknown | 0

8. Primary Outcome: Number of Participants With Hematological Abnormalities Reported as Serious Adverse Events
Description: The number of participants with hematological laboratory abnormalities reported as serious adverse events was counted. Adverse events (AEs) were encoded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 21.1. More than one serious adverse event may have been reported per participant. Participants with multiple occurrences of the same serious adverse event were only counted once per preferred term.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants | 2

9. Primary Outcome: Number of Participants With Serum Chemistry Abnormalities Reported as Serious Adverse Events
Description: The number of participants with serum chemistry laboratory abnormalities reported as serious adverse events was counted. Adverse events (AEs) were encoded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 21.1. More than one serious adverse event may have been reported per participant. Participants with multiple occurrences of the same serious adverse event were only counted once per preferred term.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants | 0

10. Primary Outcome: Number of Participants With Coagulation Abnormalities Reported as Serious Adverse Events
Description: The number of participants with coagulation laboratory abnormalities reported as serious adverse events was counted. Adverse events (AEs) were encoded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 21.1. More than one serious adverse event may have been reported per participant. Participants with multiple occurrences of the same serious adverse event were only counted once per preferred term.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants | 1

11. Primary Outcome: Number of Participants Who Died Due to a Serious Adverse Event by Cause of Death
Description: The number of participants who died due to a serious adverse event was counted by the cause of death.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Disease progression | 10
  Sepsis and disease progression | 1
  Dyspnoea | 1
  Septic shock | 1
  Shock | 1
  Unknown cause | 1

12. Primary Outcome: Overall Number of Participants by the Number of Non-Serious Adverse Events Reported Per Participant
Description: The number of participants with non-serious adverse events was counted in the four following categories for number of events reported per participant: greater than or equal to (≥) 1, 1, greater than (>) 1, or 0 non-serious adverse events. Participants with multiple occurrences of events (the ≥1 and >1 non-serious adverse event categories) were only counted once per category.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  ≥1 Non-Serious Adverse Event | 47
  1 Non-Serious Adverse Event | 11
  >1 Non-Serious Adverse Events | 36
  0 Non-Serious Adverse Events | 5

13. Primary Outcome: Overall Number of Participants With Non-Serious Adverse Events by Severity, According to NCI-CTCAE v4.03
Description: The number of participants with non-serious adverse events was counted by the severity level of the adverse event, assessed as Grades 1-5 according to NCI CTCAE v4.03. Any adverse event not specifically listed in NCI CTCAE v4.03 was assessed according to the following grades of severity: Grade 1 is mild; Grade 2 is moderate; Grade 3 is severe or medically significant; Grade 4 is life-threatening or urgent intervention indicated; and Grade 5 is death related to adverse event. The terms "severe" and "serious" are not synonymous. Severity refers to the intensity of an adverse event. The seriousness of an adverse event is based on whether it meets any of the criteria set out in the protocol's definition of a serious adverse event. Severity and seriousness were independently assessed for each adverse event. Participants with multiple occurrences of non-serious adverse events of the same severity were only counted once per severity category.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population; the number analyzed represents participants with at least one non-serious adverse event (denominator).
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Grade 1: number analyzed (Participants) | 47
  Grade 1 | 38
  Grade 2: number analyzed (Participants) | 47
  Grade 2 | 34
  Grade 3: number analyzed (Participants) | 47
  Grade 3 | 12
  Grade 4: number analyzed (Participants) | 47
  Grade 4 | 1
  Grade 5: number analyzed (Participants) | 47
  Grade 5 | 0

14. Primary Outcome: Number of Participants With Non-Serious Adverse Events Related to Docetaxel
Description: The number of participants with non-serious adverse events was counted for any non-serious adverse event that was related to study treatment with docetaxel, in the investigator's judgment. Adverse events (AEs) were encoded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 21.1. More than one non-serious adverse event may have been reported per participant. Participants with multiple occurrences of the same non-serious adverse event were only counted once per preferred term.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Any Non-Serious AEs Related to Docetaxel | 30
  Diarrhoea | 12
  Anaemia | 7
  Stomatitis | 6
  Leukopenia | 4
  Alopecia | 4
  Vomiting | 4
  Pain | 4
  Fatigue | 4
  Oedema peripheral | 3
  Skin ulcer | 2
  Hypokalaemia | 2
  Lacrimation increased | 2
  Asthenia | 2
  Pyrexia | 2
  Paraesthesia | 2
  Peripheral sensory neuropathy | 2
  Dry skin | 2
  Rash | 2
  Skin exfoliation | 2
  Muscular weakness | 1
  Febrile neutropenia | 1
  Thrombocytopenia | 1
  Sinus tachycardia | 1
  Abdominal pain | 1
  Anal fistula | 1
  Anorectal discomfort | 1
  Constipation | 1
  Frequent bowel movements | 1
  Gastritis | 1
  Haemorrhoidal haemorrhage | 1
  Hyperchlorhydria | 1
  Oral discomfort | 1
  Chest pain | 1
  Peripheral swelling | 1
  Genital herpes | 1
  Pyoderma | 1
  Skin infection | 1
  Urinary tract infection | 1
  Liver function test abnormal | 1
  Decreased appetite | 1
  Hypomagnesaemia | 1
  Hypophosphataemia | 1
  Joint swelling | 1
  Limb discomfort | 1
  Pain in extremity | 1
  Burning sensation | 1
  Neuropathy peripheral | 1
  Productive cough | 1
  Dermatitis acneiform | 1
  Rash maculo-papular | 1
  Seborrhoeic dermatitis | 1
  Skin hypertrophy | 1
  Stevens-Johnson syndrome | 1

15. Primary Outcome: Number of Participants With Non-Serious Adverse Events Related to Pertuzumab
Description: The number of participants with non-serious adverse events was counted for any non-serious adverse event that was related to study treatment with pertuzumab, in the investigator's judgment. Adverse events (AEs) were encoded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 21.1. More than one non-serious adverse event may have been reported per participant. Participants with multiple occurrences of the same non-serious adverse event were only counted once per preferred term.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Any Non-Serious AEs Related to Pertuzumab | 20
  Diarrhoea | 10
  Stomatitis | 5
  Pain | 3
  Ejection fraction decreased | 3
  Rash | 3
  Lacrimation increased | 2
  Chills | 2
  Nasal dryness | 2
  Dry skin | 2
  Oedema peripheral | 1
  Skin ulcer | 1
  Left ventricular dysfunction | 1
  Sinus tachycardia | 1
  Abdominal discomfort | 1
  Generalised oedema | 1
  Pyrexia | 1
  Hypokalaemia | 1
  Hypomagnesaemia | 1
  Myalgia | 1
  Burning sensation | 1
  Neuropathy peripheral | 1
  Breast discomfort | 1
  Productive cough | 1
  Dermatitis acneiform | 1
  Onycholysis | 1
  Rash maculo-papular | 1

16. Primary Outcome: Number of Participants With Non-Serious Adverse Events Related to Trastuzumab
Description: The number of participants with non-serious adverse events was counted for any non-serious adverse event that was related to study treatment with trastuzumab, in the investigator's judgment. Adverse events (AEs) were encoded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 21.1. More than one non-serious adverse event may have been reported per participant. Participants with multiple occurrences of the same non-serious adverse event were only counted once per preferred term.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants | 0

17. Primary Outcome: Overall Number of Participants With Non-Serious Adverse Events by Chemotherapy Adjustment With Docetaxel and/or Trastuzumab
Description: The number of participants with non-serious adverse events was counted by the type of action taken with docetaxel and/or trastuzumab in response to the adverse event in the three following categories: no adjustment, dosage modified/interrupted, and discontinued. More than one non-serious adverse event may have been reported per participant. Participants with multiple occurrences of non-serious adverse events that required the same action to be taken with the study drug were only counted once per category.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  No Adjustment: number analyzed (Participants) | 47
  No Adjustment | 45
  Dosage Modified / Interrupted: number analyzed (Participants) | 47
  Dosage Modified / Interrupted | 9
  Discontinued: number analyzed (Participants) | 47
  Discontinued | 7

18. Primary Outcome: Overall Number of Participants With Non-Serious Adverse Events by Action Taken With Pertuzumab
Description: The number of participants with non-serious adverse events was counted by the type of action taken with pertuzumab in response to the adverse event in the three following categories: no action taken, infusion slow down, infusion interrupted, and appropriate medical therapies administered. More than one non-serious adverse event may have been reported per participant. Participants with multiple occurrences of non-serious adverse events that required the same action to be taken with the study drug were only counted once per category.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  No Action Taken: number analyzed (Participants) | 47
  No Action Taken | 47
  Infusion Slow Down: number analyzed (Participants) | 47
  Infusion Slow Down | 0
  Infusion Interrupted: number analyzed (Participants) | 47
  Infusion Interrupted | 0
  Appropriate Medical Therapies Administered: number analyzed (Participants) | 47
  Appropriate Medical Therapies Administered | 0

19. Primary Outcome: Overall Number of Participants With Non-Serious Adverse Events by Event Outcome
Description: The number of participants with non-serious adverse events was counted by the event outcome in the four following categories: resolved with no sequelae, resolved with sequelae, unresolved, or death. More than one non-serious adverse event may have been reported per participant. Participants with multiple occurrences of non-serious adverse events with the same outcome were only counted once per category.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Resolved with No Sequelae: number analyzed (Participants) | 47
  Resolved with No Sequelae | 42
  Resolved with Sequelae: number analyzed (Participants) | 47
  Resolved with Sequelae | 12
  Unresolved: number analyzed (Participants) | 47
  Unresolved | 27
  Death: number analyzed (Participants) | 47
  Death | 2

20. Primary Outcome: Overall Number of Participants With Non-Serious Adverse Events by Treatment Emergence (TEAE Versus Non-TEAE)
Description: The number of participants with non-serious adverse events was counted according to whether the event was considered a treatment emergent adverse event (TEAE), which is defined as an adverse event that emerges during treatment, having been absent pretreatment, or worsens relative to the pretreatment state. Participants with multiple occurrences of non-serious adverse events were only counted once per category.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  TEAEs | 47
  Non-TEAEs | 3

21. Primary Outcome: Number of Participants With Hematological Abnormalities Reported as Non-Serious Adverse Events
Description: The number of participants with hematological laboratory abnormalities reported as non-serious adverse events was counted. Adverse events (AEs) were encoded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 21.1. More than one non-serious adverse event may have been reported per participant. Participants with multiple occurrences of the same non-serious adverse event were only counted once per preferred term.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Anaemia | 8
  Leukopenia | 4
  Neutropenia | 2
  Febrile neutropenia | 1
  Iron deficiency | 1
  Thrombocytopenia | 1

22. Primary Outcome: Number of Participants With Serum Chemistry Abnormalities Reported as Non-Serious Adverse Events
Description: The number of participants with serum chemistry laboratory abnormalities reported as non-serious adverse events was counted. Adverse events (AEs) were encoded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 21.1. More than one non-serious adverse event may have been reported per participant. Participants with multiple occurrences of the same non-serious adverse event were only counted once per preferred term.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Hypomagnesaemia | 4
  Hypokalaemia | 2
  Hypoalbuminaemia | 1
  Hypophosphataemia | 1
  Hyperglycaemia | 1
  Hyperuricaemia | 1
  Liver function test abnormal | 1

23. Primary Outcome: Number of Participants With Coagulation Abnormalities Reported as Non-Serious Adverse Events
Description: The number of participants with coagulation laboratory abnormalities reported as non-serious adverse events was counted. Adverse events (AEs) were encoded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 21.1. More than one non-serious adverse event may have been reported per participant. Participants with multiple occurrences of the same non-serious adverse event were only counted once per preferred term.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Thrombocytopenia | 1
  Anal haemorrhage | 1
  Haemorrhoidal haemorrhage | 1
  Rectal haemorrhage | 1
  Upper gastrointestinal haemorrhage | 1
  Vaginal haemorrhage | 1
  Thrombophlebitis | 1

24. Primary Outcome: Number of Participants With Congestive Heart Failure
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants | 0

25. Primary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) Over Time
Description: Left ventricular ejection fraction (LVEF) assessments were performed within 42 days of enrollment and every three treatment cycles by either echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan; ECHO was the preferred method. In order to be eligible for this study, an LVEF of ≥50% was required at screening. The same method of LVEF assessment for each participant must have been used throughout the study, and to the extent possible, have been obtained at the same institution.
Time Frame: Baseline, every 3 cycles (1 cycle is 21 days) until treatment discontinuation, at Safety Follow-Up (28 days after last dose of study drug) and every 3 months thereafter until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: percentage points of LVEF
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
percentage points of LVEF
  Baseline (BL) - Value at Visit | 59.6 (3.92)
  Change from BL at Cycle 3: number analyzed (Participants) | 51
  Change from BL at Cycle 3 | -0.7 (2.95)
  Change from BL at Cycle 6: number analyzed (Participants) | 40
  Change from BL at Cycle 6 | -0.8 (4.09)
  Change from BL at Cycle 9: number analyzed (Participants) | 26
  Change from BL at Cycle 9 | -0.2 (4.43)
  Change from BL at Cycle 12: number analyzed (Participants) | 17
  Change from BL at Cycle 12 | 0.2 (3.99)
  Change from BL at Cycle 15: number analyzed (Participants) | 18
  Change from BL at Cycle 15 | -0.8 (4.33)
  Change from BL at Cycle 18: number analyzed (Participants) | 13
  Change from BL at Cycle 18 | -1.3 (4.07)
  Change from BL at Cycle 21: number analyzed (Participants) | 12
  Change from BL at Cycle 21 | -1.8 (5.72)
  Change from BL at Cycle 24: number analyzed (Participants) | 9
  Change from BL at Cycle 24 | -0.7 (4.03)
  Change from BL at Cycle 27: number analyzed (Participants) | 7
  Change from BL at Cycle 27 | 0.0 (2.83)
  Change from BL at Cycle 30: number analyzed (Participants) | 4
  Change from BL at Cycle 30 | -1.3 (6.55)
  Change from BL at Cycle 33: number analyzed (Participants) | 6
  Change from BL at Cycle 33 | -0.5 (3.21)
  Change from BL at Cycle 36: number analyzed (Participants) | 6
  Change from BL at Cycle 36 | 0.0 (2.90)
  Change from BL at Cycle 39: number analyzed (Participants) | 3
  Change from BL at Cycle 39 | -1.3 (3.51)
  Change from BL at Cycle 42: number analyzed (Participants) | 2
  Change from BL at Cycle 42 | 1.0 (0)
  Change from BL at Cycle 45: number analyzed (Participants) | 2
  Change from BL at Cycle 45 | 0.0 (1.41)
  Change from BL at Cycle 48: number analyzed (Participants) | 2
  Change from BL at Cycle 48 | -2.0 (2.83)
  Change from BL at Cycle 51: number analyzed (Participants) | 1
  Change from BL at Cycle 51 | -18.0 (NA) — Standard deviation could not be calculated for a value from a single participant.
  Change from BL at Safety Follow-Up: number analyzed (Participants) | 28
  Change from BL at Safety Follow-Up | -4.3 (12.98)
  Change from BL at 3 Month Follow-Up: number analyzed (Participants) | 20
  Change from BL at 3 Month Follow-Up | -2.1 (4.80)
  Change from BL at 6 Month Follow-Up: number analyzed (Participants) | 18
  Change from BL at 6 Month Follow-Up | -1.8 (4.41)
  Change from BL at 9 Month Follow-Up: number analyzed (Participants) | 14
  Change from BL at 9 Month Follow-Up | -3.4 (6.44)
  Change from BL at 12 Month Follow-Up: number analyzed (Participants) | 10
  Change from BL at 12 Month Follow-Up | -2.3 (4.40)
  Change from BL at 15 Month Follow-Up: number analyzed (Participants) | 3
  Change from BL at 15 Month Follow-Up | -4.7 (5.51)
  Change from BL at 18 Month Follow-Up: number analyzed (Participants) | 2
  Change from BL at 18 Month Follow-Up | -10.0 (7.07)
  Change from BL at 21 Month Follow-Up: number analyzed (Participants) | 1
  Change from BL at 21 Month Follow-Up | -5.0 (NA) — Standard deviation could not be calculated for a value from a single participant.
  Change from BL at 24 Month Follow-Up: number analyzed (Participants) | 1
  Change from BL at 24 Month Follow-Up | -5.0 (NA) — Standard deviation could not be calculated for a value from a single participant.

26. Primary Outcome: Number of Participants by Left Ventricular Ejection Fraction (LVEF) Findings Over Time
Description: Left ventricular ejection fraction (LVEF) assessments were performed within 42 days of enrollment and every three treatment cycles by either echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan; ECHO was the preferred method. In order to be eligible for this study, an LVEF greater than or equal to (≥)50% was required at screening. The same method of LVEF assessment for each participant must have been used throughout the study, and to the extent possible, have been obtained at the same institution. The following are definitions for the three categories of LVEF findings: 'Normal' was defined as LVEF ≥45%; 'Abnormal but not clinically significant' was defined as LVEF <45% but not clinically significant in the investigator's judgment; 'Abnormal and clinically significant' was defined as LVEF <45% and clinically significant in the investigator's judgment.
Time Frame: as for outcome 25
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Baseline: Normal | 50
  Baseline: Abnormal But Not Clinically Significant | 2
  Baseline: Abnormal and Clinically Significant | 0
  Cycle 3: number analyzed (Participants) | 51
  Cycle 3: Normal | 48
  Cycle 3: Abnormal But Not Clinically Significant | 3
  Cycle 3: Abnormal and Clinically Significant | 0
  Cycle 6: number analyzed (Participants) | 40
  Cycle 6: Normal | 37
  Cycle 6: Abnormal But Not Clinically Significant | 3
  Cycle 6: Abnormal and Clinically Significant | 0
  Cycle 9: number analyzed (Participants) | 26
  Cycle 9: Normal | 24
  Cycle 9: Abnormal But Not Clinically Significant | 1
  Cycle 9: Abnormal and Clinically Significant | 1
  Cycle 12: number analyzed (Participants) | 17
  Cycle 12: Normal | 17
  Cycle 12: Abnormal But Not Clinically Significant | 0
  Cycle 12: Abnormal and Clinically Significant | 0
  Cycle 15: number analyzed (Participants) | 18
  Cycle 15: Normal | 16
  Cycle 15: Abnormal But Not Clinically Significant | 2
  Cycle 15: Abnormal and Clinically Significant | 0
  Cycle 18: number analyzed (Participants) | 13
  Cycle 18: Normal | 11
  Cycle 18: Abnormal But Not Clinically Significant | 2
  Cycle 18: Abnormal and Clinically Significant | 0
  Cycle 21: number analyzed (Participants) | 12
  Cycle 21: Normal | 10
  Cycle 21: Abnormal But Not Clinically Significant | 1
  Cycle 21: Abnormal and Clinically Significant | 1
  Cycle 24: number analyzed (Participants) | 9
  Cycle 24: Normal | 8
  Cycle 24: Abnormal But Not Clinically Significant | 1
  Cycle 24: Abnormal and Clinically Significant | 0
  Cycle 27: number analyzed (Participants) | 7
  Cycle 27: Normal | 5
  Cycle 27: Abnormal But Not Clinically Significant | 2
  Cycle 27: Abnormal and Clinically Significant | 0
  Cycle 30: number analyzed (Participants) | 4
  Cycle 30: Normal | 3
  Cycle 30: Abnormal But Not Clinically Significant | 1
  Cycle 30: Abnormal and Clinically Significant | 0
  Cycle 33: number analyzed (Participants) | 6
  Cycle 33: Normal | 5
  Cycle 33: Abnormal But Not Clinically Significant | 1
  Cycle 33: Abnormal and Clinically Significant | 0
  Cycle 36: number analyzed (Participants) | 6
  Cycle 36: Normal | 5
  Cycle 36: Abnormal But Not Clinically Significant | 1
  Cycle 36: Abnormal and Clinically Significant | 0
  Cycle 39: number analyzed (Participants) | 3
  Cycle 39: Normal | 2
  Cycle 39: Abnormal But Not Clinically Significant | 1
  Cycle 39: Abnormal and Clinically Significant | 0
  Cycle 42: number analyzed (Participants) | 2
  Cycle 42: Normal | 2
  Cycle 42: Abnormal But Not Clinically Significant | 0
  Cycle 42: Abnormal and Clinically Significant | 0
  Cycle 45: number analyzed (Participants) | 2
  Cycle 45: Normal | 2
  Cycle 45: Abnormal But Not Clinically Significant | 0
  Cycle 45: Abnormal and Clinically Significant | 0
  Cycle 48: number analyzed (Participants) | 2
  Cycle 48: Normal | 2
  Cycle 48: Abnormal But Not Clinically Significant | 0
  Cycle 48: Abnormal and Clinically Significant | 0
  Cycle 51: number analyzed (Participants) | 1
  Cycle 51: Normal | 0
  Cycle 51: Abnormal But Not Clinically Significant | 0
  Cycle 51: Abnormal and Clinically Significant | 1
  Safety Follow-Up: number analyzed (Participants) | 28
  Safety Follow-Up: Normal | 24
  Safety Follow-Up: Abnormal But Not Clinically Significant | 1
  Safety Follow-Up: Abnormal and Clinically Significant | 3
  3 Month Follow-Up: number analyzed (Participants) | 20
  3 Month Follow-Up: Normal | 17
  3 Month Follow-Up: Abnormal But Not Clinically Significant | 3
  3 Month Follow-Up: Abnormal and Clinically Significant | 0
  6 Month Follow-Up: number analyzed (Participants) | 18
  6 Month Follow-Up: Normal | 18
  6 Month Follow-Up: Abnormal But Not Clinically Significant | 0
  6 Month Follow-Up: Abnormal and Clinically Significant | 0
  9 Month Follow-Up: number analyzed (Participants) | 14
  9 Month Follow-Up: Normal | 13
  9 Month Follow-Up: Abnormal But Not Clinically Significant | 0
  9 Month Follow-Up: Abnormal and Clinically Significant | 1
  12 Month Follow-Up: number analyzed (Participants) | 10
  12 Month Follow-Up: Normal | 10
  12 Month Follow-Up: Abnormal But Not Clinically Significant | 0
  12 Month Follow-Up: Abnormal and Clinically Significant | 0
  15 Month Follow-Up: number analyzed (Participants) | 3
  15 Month Follow-Up: Normal | 3
  15 Month Follow-Up: Abnormal But Not Clinically Significant | 0
  15 Month Follow-Up: Abnormal and Clinically Significant | 0
  18 Month Follow-Up: number analyzed (Participants) | 2
  18 Month Follow-Up: Normal | 2
  18 Month Follow-Up: Abnormal But Not Clinically Significant | 0
  18 Month Follow-Up: Abnormal and Clinically Significant | 0
  21 Month Follow-Up: number analyzed (Participants) | 1
  21 Month Follow-Up: Normal | 1
  21 Month Follow-Up: Abnormal But Not Clinically Significant | 0
  21 Month Follow-Up: Abnormal and Clinically Significant | 0
  24 Month Follow-Up: number analyzed (Participants) | 1
  24 Month Follow-Up: Normal | 1
  24 Month Follow-Up: Abnormal But Not Clinically Significant | 0
  24 Month Follow-Up: Abnormal and Clinically Significant | 0

27. Primary Outcome: Number of Participants With Adverse Events Leading to Treatment Discontinuation
Description: The number of participants with any adverse event (serious or non-serious) that led to treatment discontinuation during the study was counted. Adverse events (AEs) were encoded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 21.1. More than one adverse event that led to treatment discontinuation may have been reported per participant.
Time Frame: From Baseline until end of study (up to approximately 3 years)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Any AEs Leading to Treatment Discontinuation | 16
  Disease progression | 5
  Ejection fraction decreased | 3
  Headache | 2
  Anaemia | 1
  Death | 1
  Diarrhoea | 1
  Dyspnoea | 1
  Febrile neutropenia | 1
  Infusion related reaction | 1
  Sepsis | 1
  Septic shock | 1
  Shock | 1
  Stevens-Johnson syndrome | 1

28. Secondary Outcome: Overall Response Rate
Description: The overall response rate (ORR) was defined as the percentage of participants with best overall response of Complete Response (CR) or Partial Response (PR), confirmed by repeat assessment no less than 4 weeks after the response criteria were first met, using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). Participants who either had not achieved CR or PR or were without a post-baseline tumor assessment were to be considered non-responders. All measurable and non-measurable lesions were documented at screening and re-assessed at each subsequent tumor evaluation. Response was assessed by the investigator on the basis of physical examinations, computed tomography (CT) scans, and magnetic resonance imaging (MRI). The same radiographic procedure was used throughout the study, and assessments were preferably performed by the same evaluator. The 95% confidence intervals were calculated using Clopper-Pearson methodology.
Time Frame: From Baseline up to disease progression or death (assessed at every 9 weeks, up to approximately 3 years)
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
percentage of participants
  Responders (ORR) | 82.7 [69.67 to 91.77]
  Non-Responders | 17.3 [8.23 to 30.33]

29. Secondary Outcome: Number of Participants by Best Overall Response
Description: The best overall response was defined as the best response, out of all the documented responses over the course of the entire study period, using RECIST v1.1. All measurable and non-measurable lesions were documented at screening and re-assessed at each subsequent tumor evaluation. Response was assessed by the investigator on the basis of physical examinations, computed tomography (CT) scans, and magnetic resonance imaging (MRI). The same radiographic procedure was used throughout the study, and assessments were preferably performed by the same evaluator.
Time Frame: From Baseline up to disease progression or death (assessed at every 9 weeks, up to approximately 3 years)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 43
  Progressive Disease (PD) | 1
  Stable Disease (SD) | 6
  Unable to Assess | 2

30. Secondary Outcome: Number of Participants With Disease Progression or Death or Who Were Censored for Progression-Free Survival Analysis
Description: Progression-free survival (PFS) was defined as the time from enrollment to the first occurrence of disease progression as determined by the investigator using RECIST v1.1, or death from any cause, whichever occurred first. Participants who had not progressed or died or were lost to follow up at the time of the analysis were censored on the last visit at which assessment for progression was done (2 years after the last participant was enrolled). PFS was analyzed by the Kaplan-Meier method.
Time Frame: From Baseline up to disease progression or death (assessed at every 9 weeks, up to approximately 3 years)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Disease Progression or Death | 32
  Censored | 20

31. Secondary Outcome: Median Duration of Progression-Free Survival
Description: Progression-free survival (PFS) was defined as the time from enrollment to the first occurrence of disease progression as determined by the investigator using RECIST v1.1, or death from any cause, whichever occurred first. Participants who had not progressed or died, or were lost to follow up at the time of the analysis, were censored on the last visit at which assessment for progression was done (2 years after the last participant was enrolled). PFS was analyzed by the Kaplan-Meier method.
Time Frame: From Baseline up to disease progression or death (assessed at every 9 weeks, up to approximately 3 years)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
months | 23.0 [13.0 to 29.0]

32. Secondary Outcome: Probability of Participants Remaining Event-Free in Progression-Free Survival From 2 to 32 Months
Description: Progression-free survival (PFS) was defined as the time from enrollment to the first occurrence of disease progression as determined by the investigator using RECIST v1.1, or death from any cause, whichever occurred first. Participants who had not progressed, died or were lost to follow up at the time of the analysis were censored on the last visit at which assessment for progression was done (2 years after the last participant was enrolled). PFS was analyzed by the Kaplan-Meier method.
Time Frame: Months 2, 3, 5, 6, 7, 8, 9, 11, 13, 15, 16, 17, 18, 19, 23, 24, 25, 27, 29, and 32
Population: ITT Population
Measure: Number; unit: Percent probability of PFS
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Percent probability of PFS
  At 2 Months | 98.08
  At 3 Months | 96.15
  At 5 Months | 90.27
  At 6 Months | 88.30
  At 7 Months | 82.42
  At 8 Months | 78.49
  At 9 Months | 74.57
  At 11 Months | 68.52
  At 13 Months | 64.49
  At 15 Months | 60.33
  At 16 Months | 58.10
  At 17 Months | 55.86
  At 18 Months | 53.63
  At 19 Months | 51.30
  At 23 Months | 48.96
  At 24 Months | 46.63
  At 25 Months | 41.72
  At 27 Months | 36.16
  At 29 Months | 32.87
  At 32 Months | 29.59

33. Secondary Outcome: Number of Participants Who Died or Were Censored for Overall Survival Analysis
Description: Overall survival was defined as the time from enrollment to the the date of death from any cause. Participants who were alive at the time of the analysis, dropped out of the study, or lost to follow-up were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last study medication, and participants with no post-baseline information were censored at baseline. Overall survival was analyzed by the Kaplan-Meier method.
Time Frame: From Baseline up to death from any cause (up to approximately 3 years)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Participants
  Death | 15
  Censored | 37

34. Secondary Outcome: Median Duration of Overall Survival
Description: as for outcome 33
Time Frame: From Baseline up to death from any cause (up to approximately 3 years)
Population: ITT Population
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
months | NA [26 to NA] — The median and the upper limit of the inter-quartile range of OS duration were not estimable because they were not reached at the time of analysis.

35. Secondary Outcome: Probability of Participants Remaining Alive in Overall Survival From 3 to 34 Months
Description: as for outcome 33
Time Frame: Months 3, 9, 13, 14, 15, 18, 19, 20, 24, 25, 27, 32, 33, and 34
Population: ITT Population
Measure: Number; unit: Percent probability of OS
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
Number analyzed (Participants) | 52
Percent probability of OS
  At 3 Months | 96.15
  At 9 Months | 88.30
  At 13 Months | 88.30
  At 14 Months | 88.30
  At 15 Months | 88.30
  At 18 Months | 83.66
  At 19 Months | 83.66
  At 20 Months | 83.66
  At 24 Months | 81.12
  At 25 Months | 81.12
  At 27 Months | 68.14
  At 32 Months | 68.14
  At 33 Months | 64.36
  At 34 Months | 64.36

ADVERSE EVENTS:
Time Frame: From Baseline until end of study (up to 3 years)
Description: After informed consent, and prior to dosing, serious adverse events (SAEs) considered related to a study mandated procedure were reportable. As of cycle 1 all adverse events and SAEs were monitored continuously and collected until the end-of-study visit.
Arm/Group | Pertuzumab in Combination With Trastuzumab and Docetaxel
All-Cause Mortality (participants affected / at risk) | 15/52
Serious Adverse Events (participants affected / at risk) | 31/52
Other Adverse Events (participants affected / at risk) | 47/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pertuzumab in Combination With Trastuzumab and Docetaxel (N=52)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Death (General disorders) | 3 (3)
Disease progression (General disorders) | 6 (6)
Fatigue (General disorders) | 3 (3)
Multiple organ dysfunction syndrome (General disorders) | 2 (2)
Septic shock (Infections and infestations) | 2 (2)
Ejection fraction decreased (Investigations) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Congenital arterial malformation (Congenital, familial and genetic disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Osteomyelitis salmonella (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pertuzumab in Combination With Trastuzumab and Docetaxel (N=52)
Diarrhoea (Gastrointestinal disorders) | 17 (43)
Stomatitis (Gastrointestinal disorders) | 8 (13)
Anaemia (Blood and lymphatic system disorders) | 8 (11)
Pyrexia (General disorders) | 8 (10)
Leukopenia (Blood and lymphatic system disorders) | 4 (6)
Lymphoedema (Vascular disorders) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7)
Vomiting (Gastrointestinal disorders) | 6 (7)
Pain (General disorders) | 5 (7)
Nasopharyngitis (Infections and infestations) | 5 (7)
Oedema peripheral (General disorders) | 4 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (6)
Lacrimation increased (Eye disorders) | 5 (6)
Headache (Nervous system disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (13)
Dizziness (Nervous system disorders) | 6 (7)
Fatigue (General disorders) | 8 (8)
Asthenia (General disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Chills (General disorders) | 4 (4)
Peripheral swelling (General disorders) | 3 (4)
Viral infection (Infections and infestations) | 3 (4)
Ejection fraction decreased (Investigations) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Paraesthesia (Nervous system disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 2 (3)
Pericardial effusion (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 2 (2)
Anal fistula (Gastrointestinal disorders) | 1 (3)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1)
Anal inflammation (Gastrointestinal disorders) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 1 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (3)
Disease progression (General disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1)
Carbuncle (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 2 (2)
Furuncle (Infections and infestations) | 1 (1)
Genital herpes (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Lymph gland infection (Infections and infestations) | 1 (1)
Pyoderma (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 1 (2)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Meibomianitis (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Breast procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Burning sensation (Nervous system disorders) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Speech disorder developmental (Nervous system disorders) | 1 (1)
Breast discomfort (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (2)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (4)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2014-06-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT02445586/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT02445586/SAP_001.pdf